CLINICAL TRIAL: NCT04766450
Title: Effect of High-Dose N-acetyl Cysteine (NAC) on the Inflammatory Markers and Clinical Outcome of Patients With Diabetic Peripheral Neuropathy (DPN)
Brief Title: Effect of High-Dose NAC on Patients With DPN
Acronym: NAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sherien Emara, Teaching Assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAC in DPN
Record Dates: First submitted 2021-02-13; First posted 2021-02-23 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1, NAC group (Active Comparator): Group 1, NAC group (n=30): Patients will receive conventional therapy for diabetic neuropathy in addition to High Dose N-acetyl cysteine (2400 mg/day divided into two doses) daily for 3 months
  Interventions: Drug: Acetyl cysteine
- Group 2, Control group (No Intervention): Group 2, Control group (n= 30): Patients will receive conventional therapy for diabetic neuropathy alone for 3 months.

INTERVENTIONS:
Drug: Acetyl cysteine — NAC exhibits potent anti-oxidant activity in the cell through augmentation of intracellular GSH, which is a major component of the pathways by which cells are protected from OTS, and its direct scavenging activity of free radicals by providing sulfhydryl groups. Additionally, NAC treatment exhibits anti-inﬂammatory effects via inhibition of NF-κB activation and reducing subsequent cytokine production . Mitochondria-protective mechanisms of NAC may also be related to its anti-oxidant and anti-inﬂammatory properties
  Other Names: N-acetyl cysteine
  Arms: Group 1, NAC group

SUMMARY:
The aim of the current study is to evaluate the efficacy and safety of high dose oral NAC (2400 mg/day divided into two doses) as an adjunct therapy on oxidative stress, inflammatory markers and clinical outcome in patients with type 2 diabetes suffering from diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Patient written informed consent will be taken prior to study conductance

* Lab assessment will be done at baseline and at the end of the study by withdrawing 7 ml of whole blood for assessment of following parameters: HbA1c, Liver & renal functions
* Inflammatory markers including: Human Nuclear factor erythroid 2-related factor (NRF2) & Tumor necrosis factor alpha (TNF-α) using ELISA Kit
* Oxidative stress markers: Glutathione Peroxidase using ELISA Kit

Inflammatory and oxidative stress marker samples will be stored at -80 for further evaluation using ELISA kit at the end of the study

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18-50 years diagnosed with Type 2 Diabetes taking oral hypoglycemic with controlled at HbA1c (6%-7%.)
2. Patients diagnosed with Diabetic Neuropathy (by pinprick, temperature probe, ankle reflex, and vibration perception (128-Hz tuning fork) or pressure sensation (10 g monofilament test).

Exclusion Criteria:

1. Patients with acute and chronic inflammatory conditions, consuming any antioxidant supplements or anti-inflammatory medicines.
2. Pregnancy or lactation or expecting to get pregnant during the study.
3. Medical, psychological, or pharmacological factors interfering with the collection or interpretation of study data.
4. Cancer patients.
5. Anyone having hypersensitivity to N-acetylcysteine.
6. Anyone already taking N-acetylcysteine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of Human Nuclear factor erythroid 2-related factor (NRF2) | change from baseline Human Nuclear factor erythroid 2-related factor at 3 months
  Inflammatory marker
Concentration of Tumor necrosis factor alpha | Change from baseline tumor necrosis factor alpha at 3 months
  Inflammatory marker
Concentration of Glutathione peroxidase | Change from baseline glutathione peroxidase at 3 months
  Oxidative stress markers

OTHER OUTCOMES:
Michigan neuropathy screening instrument. | At baseline and after 3 months
  Questionnaire of 15 yes or no questions. score of 13 or more means more neuropathic symptoms
Toronto clinical scoring system | At baseline and after 3 months
  Questionnaire. as score increase means symptoms increase

CONTACTS AND LOCATIONS:
Overall Officials: Lamia El Wakeel, Professor, Study Director — Ain Shams University
Locations (1):
- Demerdash Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Emara SM, Fahmy SF, AbdelSalam MM, Wakeel LME. Effect of high-dose N-acetyl cysteine on the clinical outcome of patients with diabetic peripheral neuropathy: a randomized controlled study. Diabetol Metab Syndr. 2025 Mar 4;17(1):79. doi: 10.1186/s13098-025-01624-9. PMID 40038825
- See also: Berk, M., Malhi, G. S., Gray, L. J., & Dean, O. M. (2013). The promise of N-acetylcysteine in neuropsychiatry. Trends in Pharmacological Sciences, 34(3), 167-177. — https://doi.org/10.1016/j.tips.2013.01.001